CLINICAL TRIAL: NCT06236035
Title: Intraoperative Analgesia Management by Monitoring Analgesia Nociception Index (ANI) in Total Knee Arthroplasty With Femoral Nerve Block: a Randomized Controlled Study
Brief Title: Intraoperative Analgesia Based on ANI
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Keziban Bollucuoglu, Principal Investigator, Zonguldak Bulent Ecevit University
Other Study IDs: 2022/04-21
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Pain Monitoring; Pain Assessment; Opioid Consumption
Keywords: Analgesia nociception index; opioid consumption; Pain management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Control
- Group ANI
  Interventions: Device: Analgesia nociception index

INTERVENTIONS:
Device: Analgesia nociception index — a device to assess patient's pain during surgery
  Groups: Group ANI

SUMMARY:
Osteoarthritis of the knee joint is common and total knee arthroplasty (TKA) is performed in patients with advanced joint degeneration, no response to conservative treatments, severe pain and joint instability. Severe pain levels between 4 and 8 in visual analog pain scale (VAS) scores have been reported in the postoperative period. Multimodal analgesia is considered to be the best option for pain control after total knee arthroplasty. Multimodal analgesia is defined as the combined use of different analgesia techniques such as neuraxial analgesia, peripheral nerve blocks, patient-controlled analgesia and different analgesic drugs. For this purpose, peripheral nerve blocks are effectively applied as a component of multimodal analgesia. Thus, side effects such as nausea, vomiting, pruritus and sedation that may occur due to opioid use are reduced. At the same time, in addition to providing effective analgesia, peripheral blocks contribute to early initiation of rehabilitation of the knee joint, early ambulation, reduction of pulmonary complications and early discharge from the hospital.

Recently, objective methods such as skin vasomotor reflex analysis, pupilometry, pulse plethysmographic signals and analgesia nociceptive index (ANI) have been used to standardize the need for intraoperative analgesia in patients under general anesthesia. Among these methods, ANI is a non-invasive method that provides continuous measurement of parasympathetic tone, which is a part of the autonomic nervous system. Electrodes are placed on the chest wall on both sides of the heart and the patient is monitored.

The investigators aimed to compare the analgesia nociception index (ANI) and the conventional method to determine perioperative analgesic needs in patients undergoing total knee arthroplasty under general anesthesia with femoral nerve block.

ELIGIBILITY:
Inclusion Criteria:

1.18-75 years old, 2.ASA I-II-III risk group 3.undergo knee operation under general anesthesia 4. Patients with preoperative femoral nerve block 5. Patients whose informed consent was read and consent was obtained from them and their guardian

Exclusion Criteria:

1. Those who do not want to participate in the study,
2. ASA IV-V patients
3. Those with central or autonomic nervous system disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 18-75 years old, ASA I-II-III risk group, undergo knee operation under general anesthesia
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
intraoperatively total opioid consumption | during the surgery
  total remifentanil consumption during surgery

SECONDARY OUTCOMES:
pain scores | up to 24 hours after surgery
  assessment pain scores by numeric rating scale (min:0, max:10)
postoperatif analgesic requirement | up to 24 hours after surgery
  need for analgesics after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No